CLINICAL TRIAL: NCT02051374
Title: Degenerative Lumbar Spondylolisthesis: Is Only Decompression Good Enough? A Prospective Randomized Clinical Multi- Institutional Trial
Brief Title: The NORDSTEN Study - Degenerative Spondylolisthesis
Acronym: NORDSTEN/DS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Møre og Romsdal Hospital Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013/366; 2013/366
Record Dates: First submitted 2014-01-10; First posted 2014-01-31 (Estimated); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Lumbar Degenerative Spondylolisthesis
MeSH Terms: interventions — Decompression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Decompression alone (Active Comparator): Posterior approach with decompression will be performed. The decompression will be done after microsurgical principles, and the midline structures will be preserved. The surgeons will either use microscope or magnifying glasses.
  Interventions: Procedure: Decompression alone
- Decompression followed by fusion with instrumentation (Active Comparator): Posterior approach with decompression will be performed, followed by posterolateral pedicle screw fixation with or without an additional cage. The surgeons will either use microscope or magnifying glasses.
  Interventions: Procedure: Decompression followed by fusion with instrumentation

INTERVENTIONS:
Procedure: Decompression alone
  Arms: Decompression alone
Procedure: Decompression followed by fusion with instrumentation
  Arms: Decompression followed by fusion with instrumentation

SUMMARY:
Lumbar Degenerative Spondylolisthesis (LDS) is a slippage of one vertebra over another caused by degeneration of facet joints, ligaments and intervertebral discs. Most patients suffer from symptoms related to spinal stenosis, such as radiating pain to the lower extremities, and typically increased pain in the lower limbs when walking upright and decreased when bending forward.

There is a moderate grade of evidence for whether patients will achieve better outcome after surgery when decompression is followed by fusion. In theory, fusion following decompression should give more stability to the operated level, thus less pain and less progression of the olisthesis. On the other hand, fusion procedures, in general, are associated with more severe complications and postoperative mortality than decompression alone.

In summary, there is still insufficient evidence for performing fusion in addition to decompression for patients with LDS. The investigators are planning a trial where the main aim is to detect whether the intervention-related difference in outcome between decompression alone (DA) and decompression followed by fusion with instrumentation (DF) is large enough to justify the use of the fusion procedure. The proposed trial is a randomized, controlled, multicentre, non- inferiority trial with two parallel groups, with 15 participating Norwegian hospitals. The main analysis will be performed 2 years after surgery with long-term follow-up planned at 5 and 10 years postoperatively.

DETAILED DESCRIPTION:
Purpose:

The aim of the study is to compare the efficacy of two principally different surgical methods for treating LDS and to investigate whether predictors will be associated with an intervention-related difference in outcome between the two groups.

Methods:

The Oswestry Disability Index (ODI) will be used as primary outcome measure in analyses at 2 year, 5 year and 10 year follow-up. Depending on whether the participants obtain a 30% or more ODI- improvement from before operation to follow-up, they will be dichotomized in a success group (responders) and in a non-success group (non- responders). The primary question is whether the proportion of patients with successful outcome in the DA group is not markedly less than in the DF group, at 2 years, 5 years and 10 years, respectively. Investigators have predefined the margin of "markedly less" to be δ = 0.15 (15%) which is consistent with the between- group difference Blumenthal et al used in the power analysis in a similar Food and Drug Administration- regulated non- inferiority RCT. With this margin it will be necessary to treat 6.7 patients with fusion in addition to decompression in order to obtain one patient with successful outcome.

The null hypothesis is that the proportion of patients with a successful outcome in the DF group (nDF) is higher than the proportion in the DA group (nDA) by an amount of at least 0.15 (δ):

H0: nDF >= nDA + δ

H0 will be tested by forming a 95% CI for the difference of proportions and H0 will be rejected if the upper limit of the confidence interval (CI) is less than 0.15.

By rejecting H0, the alternative hypothesis will be accepted:

H1: nDF < nDA + δ

By accepting H1, the conclusion will be that DA is non-inferior DF and hence as good as DF.

In addition to the efficacy analyses (main analyses)we aim to investigate the following:

I. Whether baseline parameters are associated with clinical outcomes,and whether treatment effect modifiers can be identified at the defined follow-ups (at 2 years, 5 years and 10 years) from the following list of variables:

1. Treatment group
2. Patient age
3. Gender
4. Comorbidity (ASA group)
5. Body Mass Index
6. Smoking
7. Preoperative ODI score
8. Preoperative NRS back pain
9. Preoperative NRS leg pain
10. Hopkins symptom check list (HSCL-25)
11. The magnitude of olistheses and local kyphosis measured on standing x-rays
12. Segmental instability verified on flexion/extension x-rays
13. Presence of foraminal stenosis in the level of olisthesis
14. Orientation of the facet joint in the level of olisthesis
15. Amount of facet joint fluid in the level of olisthesis
16. Degree of disc degeneration in the level of olisthesis
17. Disc height in the level of olisthesis
18. Pelvic incidence

II. Whether the surgeon's preference for treatment before randomization is associated with clinical outcomes at follow-up (2-year, 5-year and 10 year). In this study, we will use the similar primary and secondary outcome measures as for the efficacy study.

III. Health-economic comparison of decompression alone and decompression with fusion at 2-, 5- and 10-year follow-up. Details for the analysis of data up to 5-year follow-up are provided in the uploaded "Statistical Analysis Plan, NORDSTEN-DS"

This will be published in separate articles.

Sample size:

The sample size calculation is based on the hypothesis that the 2-year results for the DA group is as least as good as for the DF group when comparing the proportions of responders in each group. The sample size is computing by using the Blackwelder methodology. Based on data from the Norwegian Spine Register, the proportion of responders for the whole treatment group is expected to be 0.70. Choosing a type 1 error = 0.05, power = 0.80 and δ = 0.15 gives a sample size of 116. Considering these assumptions and adding 10% for possible dropouts, a total of 128 patients are required in each group. Using Multiple Imputation for missing data, we consider power acceptable even with some higher dropouts at 5- and 10-year follow-up.

Protocol deviations

The patients have major deviations from protocol if they:

Have not received operative treatment in accordance with randomized allocation; Have received operative treatment in accordance with randomized allocation and operated with a new operation at same level during the follow-up period; Have not provided informed consent; Have withdrew the informed consent and claimed their data withdrawn from analyses.

According to deviations to protocol the following analysis sets are defined:

Full Analysis Set (FAS): all randomised patients with primary operation according to the randomly assigned study treatment and with data on the primary outcome variable (ODI) at one or more time point.

Per Protocol Set (PPS): All randomized patients without major deviations from protocol and with data on the primary outcome variable at baseline and two-year follow-up . For 5- and 10-year analyses data are required at baseline and at the respective follow-ups.

Statistical analysis:

To determine whether randomization is successful descriptive statistics will be used for comparing baseline characteristics between the groups.

Differences in responder rates for ODI, ZCQ and NRS for leg/back pain(proportions of patients dicothomized into 'success'), including the Newcombe hybrid score confidence interval, will be estimated and tested according to non-inferiority. If there are patients with missing data at two-year follow-up, Multiple imputation (MI) will be performed including plausible baseline data and follow-up data as explanatory variables in the imputation model.

Statistical analyses will be performed both on a Full Analysis Set (FAS-MI) and a Per Protocol Set (PPS) at two-year follow-up. In the FAS-MI set missing scores necessary for dichotomizing patients into responders/non-responders will be imputed by use of Multiple imputation (MI). To recommend DA both the FAS-MI and the PPS analysis of the primary outcome are required to show non-inferiority. In addition we will perform two sensitivity analyses. One with responder analysis of FAS without imputation (a complete cases analysis) and one with responder analysis of FAS, where missing values will be replaced with values at one year follow-up, if available.

Categorical secondary outcomes will be analyzed with Fisher mid-P tests and Newcombe hybrid score intervals. The GPE responses will be analyzed with a proportional odds logistic regression model.

It will be used a linear mixed model analysis to evaluate the continous secondary outcomes, and to evaluate the effect of each efficacy variable over time and between groups (all follow-up measurements from inclusion to follow-ups will be included). In the mixed model patients are not excluded from the analysis of an efficacy variable if the variable is missing at some, but not all time points after baseline.

A significance level of 5% will be used throughout.

Data will be inaccessible to the research group until all available two-year follow-up participants has completed the 2-year questionnaire, and the study is declared adequate monitored according to principles of Good Clinical Practice (GCP).The data collected between 2- and 5-year follow up will be inaccessible to the research group until all available 5-year follow-up participants has completed the 5-year questionnaire.The data collected between 5- and 10-year follow up will be inaccessible to the research group until all available 10-year follow-up participants has completed the 10-year questionnaire.. Faculty of Research support, University of Oslo will declare this inaccessibleness and state which date the data has been accessible for the investigators.

Interim analysis and stopping rules:

When 75 patients in each group have completed the 12 months follow- up, the investigators will do an interim analysis. Due to ethical considerations the inclusion of patients will be terminated if the analysis reveals one of the following:

1. The proportion of patients with successful outcome in the DF group is higher than in the DA group by an amount of 0.20.
2. The proportion of patients needing reoperation due to any condition in the operated level(s) is statistically significant higher in one of the groups.

The interim analysis was conducted on February 28, 2017 by an independent statistician blinded for treatment adherence. Only data on reoperations and on the primary outcome measure (ODI) was available to the statistician. None of the stop criteria were fulfilled. The statistician informed the steering committee, via the central coordinator, that the study could be continued. Further information about the analysis was not disclosed and will not be available to anyone until the main analysis of 2-year follow-up data.

The reporting of the trial will be based on an adapted Consolidated Standards of Reporting Trials (CONSORT) checklist for reporting non- inferiority trials.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* do understand Norwegian language, spoken and in writing
* have a degenerative lumbar spondylolisthesis, with a slip >=3 mm, verified on standing plain x-rays in lateral view
* have a spinal stenosis in the level of spondylolisthesis, shown on MRI
* have clinical symptoms of spinal stenosis as neurogenic claudication or radiating pain into the lower limbs, not responding to at least 3 months of qualified conservative treatment
* are able to give informed consent and to respond to the questionnaires.

Exclusion Criteria:

* are not willing to give written consent
* are participating in another clinical trial that may interfere with this trial
* are ASA- classified > 3
* are older than 80 years
* are not able to comply fully with the protocol, including treatment, follow-up or study procedures (psychosocially, mentally and physical)
* have cauda equina syndrome (bowel or bladder dysfunction) or fixed complete motor deficit
* have a slip >=3 mm in more than one level
* have an isthmic defect in pars interarticularis
* have a fracture or former fusion of the thoracolumbal region
* have had previous surgery in the level of spondylolisthesis
* have a lumbosacral scoliosis more than 20 degrees verified on AP-view
* have distinct symptoms in one or both legs due to other diseases, e.g. polyneuropathy, vascular claudication or osteoarthritis
* have radicular pain due to a MRI verified foraminal stenosis in the slipped level, with deformation of the nerve root because of a bony narrowing in the vertical direction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
The Oswestry Disability Index | Prior to operation and 3 months, 1 year, 2 years, 5 years and 10 years postoperatively.
  The Oswestry Disability Index (ODI) version 2.0 will be used as primary outcome measure. ODI is widely used by physicians treating patients with back-related symptoms and has been translated and validated for applications with Norwegian patients. It is a self-reported instrument comprising 10 sections where the patient is supposed to mark the most appropriate item. ODI scores range from 0 to 100, where 100 is the greatest impairment.
  The percentage change in ODI from baseline to follow- up will be computed. An individual cutoff value of 30% ODI- improvement will be used to dichotomize the patients in a success group and in a non- success group. This threshold value is estimated based on data from patients registered in the Norwegian registry for Spine Surgery The change in ODI from before operation to follow up will also be computed and reported as means.

SECONDARY OUTCOMES:
Zürich Claudication Questionnaire (ZCQ): | Prior to operation and 3 months, 1 year, 2 years, 5 years and 10 years postoperatively.
  Zürich Claudication Questionnaire is also known as the Swiss Spinal Stenosis Questionaire, and is a self-completed disorder-specific functional score consisting of three domains: symptom severity, physical function and patient satisfaction. The questionnaire is translated and validated for use on Norwegian patients suffering from degenerative lumbar spinal stenosis.
  The change in ZCQ from baseline to follow- up will be computed. An individual cutoff value will be used to dichotomize the patients in a success group and in a non- success group.
Numeric Rating Scale (NRS) for back- and leg pain | Prior to operation and 3 months, 1 year, 2 years, 5 years and 10 years postoperatively.
  NRS is a PRO that assesses self-reported pain the patients experienced in the last week from 0 (no pain) to 10 (the worst pain imaginable), on a horizontal 10 centimeter scale. The change in NRS from baseline to follow- up will be computed separately for leg and back pain.Based on data from NORSpine, the individual thresholds for being a responder are defined as a 40% reduction in the NRS leg pain and a 33% reduction in NRS back pain.
Euroquol 5 dimensions questionnaire (EQ-5D) | Prior to operation, 3 months, 1 year, 2 years, 5 years and 10 years postoperatively.
  EQ-5D is a generic PRO that is self-completed and comprises 5 questions relating to mobility, self-care, usual activity, pain/discomfort, and anxiety/depression. It is one of the most frequent used questionnaires in determining cost- effectiveness in health economic evaluation. We will consider doing such an evaluation as part of the secondary outcome analysis.
Global Perceived Effect (GPE) scale: | 3 months, 1 year, 2 years, 5 years and 10 years postoperatively.
  Patient- rated satisfaction with treatment and treatment outcome will be assessed using single question with seven-point descriptive scaling.
Percentages of participants with adverse effects (complications) | During the hospital stay (average 2-3 days) and up to 10 years postoperatively.
  A research coordinator will record complications consecutively during the hospital stay. These may include infections, hematoma, neurological deficits due to the operation, CSF leakage and other major adverse effects. Later complications such as wound infections and hardware failure, will be recorded by the self- questionnaires.
Percentages of participants needing a reoperation. | 3 months, 1 year, 2 years, 5 years and 10 years postoperatively.
  Any new operation in the primary operated level during the follow- up period will be recorded as a reoperation.
Duration of surgery | At disharge from hospital at primary operation.
  The time from opening to closing the skin
Length of hospital stay | At disharge from hospital at primary operation.
  The number of days from operation to discharge from the hosptal
Volume of blood loss and use of blood transfusion | At disharge from hospital at primary operation.
  Volume of blood loss during the operation and volum of blood transfusion during hospital stay

OTHER OUTCOMES:
Radiological findings | MRI: Prior to operation. Skeletal x-rays:Prior to operation, at 3 month follow- up and at 2 year follow- up. CT scan: At 2 year follow- up.
  Radiological parameters will be reported, but not evaluated as outcomes parameters:
  1. MRI of the lumbar spine, including T1 and T2 sequences in the axial and sagittal plane.
  2. Skeletal x-rays:
     * Standard images; frontal and lateral view of L1 to S1 in standing position.
     * Ex/flex- images; lateral view of L1 to S1 with respectively maximal flexion and maximal extension
  3. CT scan: To compute the fusion rate. "Union" is classified as bony continuity between the fused vertebrae in both the coronal and sagittal view.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Hellum, MD, PhD, Study Chair — Orthopeadic Clinic, Oslo University Hospital; Ivar Magne Austevoll, Md, PhD, Principal Investigator — Kysthospitalet i Hagevik, Orthopeadic Clinic, Haukeland University Hospital; Eric Loratang Kgomotso, MD, Principal Investigator — Kysthospitalet i Hagevik, Orthopeadic Clinic, Haukeland University Hospital
Locations (1):
- Kysthospitalet i Hagevik, Orthopeadic Clinic, Haukeland University Hospital, Bergen, Hagevik, Norway

REFERENCES:
- [Derived] Indrekvam K, Myklebust TA, Austevoll IM, Hermansen E, Banitalebi H, Banerud IF, Weber C, Brisby H, Brox JI, Hellum C, Storheim K. Responsiveness of the Oswestry Disability Index and Zurich Claudication Questionnaire in patients with lumbar spinal stenosis: evaluation of surgically treated patients from the NORDSTEN study. Eur Spine J. 2024 Nov;33(11):4270-4280. doi: 10.1007/s00586-024-08440-1. Epub 2024 Aug 13. PMID 39134699
- [Derived] Kgomotso EL, Hellum C, Fagerland MW, Solberg T, Brox JI, Storheim K, Hermansen E, Franssen E, Weber C, Brisby H, Algaard KRH, Furunes H, Banitalebi H, Ljostad I, Indrekvam K, Austevoll IM; Nordsten collaborators. Decompression alone or with fusion for degenerative lumbar spondylolisthesis (Nordsten-DS): five year follow-up of a randomised, multicentre, non-inferiority trial. BMJ. 2024 Aug 7;386:e079771. doi: 10.1136/bmj-2024-079771. PMID 39111800
- [Derived] Indrekvam K, Banerud IF, Hermansen E, Austevoll IM, Rekeland F, Guddal MH, Solberg TK, Brox JI, Hellum C, Storheim K. The Norwegian degenerative spondylolisthesis and spinal stenosis (NORDSTEN) study: study overview, organization structure and study population. Eur Spine J. 2023 Dec;32(12):4162-4173. doi: 10.1007/s00586-023-07827-w. Epub 2023 Jul 3. PMID 37395780
- [Derived] Hellum C, Rekeland F, Smastuen MC, Solberg T, Hermansen E, Storheim K, Brox JI, Furunes H, Franssen E, Weber C, Brisby H, Grundnes O, Algaard KRH, Boker T, Banitalebi H, Indrekvam K, Austevoll IM. Surgery in degenerative spondylolisthesis: does fusion improve outcome in subgroups? A secondary analysis from a randomized trial (NORDSTEN trial). Spine J. 2023 Nov;23(11):1613-1622. doi: 10.1016/j.spinee.2023.06.386. Epub 2023 Jun 22. PMID 37355044
- [Derived] Austevoll IM, Hermansen E, Fagerland MW, Storheim K, Brox JI, Solberg T, Rekeland F, Franssen E, Weber C, Brisby H, Grundnes O, Algaard KRH, Boker T, Banitalebi H, Indrekvam K, Hellum C; NORDSTEN-DS Investigators. Decompression with or without Fusion in Degenerative Lumbar Spondylolisthesis. N Engl J Med. 2021 Aug 5;385(6):526-538. doi: 10.1056/NEJMoa2100990. PMID 34347953
- [Derived] Austevoll IM, Hermansen E, Fagerland M, Rekeland F, Solberg T, Storheim K, Brox JI, Lonne G, Indrekvam K, Aaen J, Grundnes O, Hellum C. Decompression alone versus decompression with instrumental fusion the NORDSTEN degenerative spondylolisthesis trial (NORDSTEN-DS); study protocol for a randomized controlled trial. BMC Musculoskelet Disord. 2019 Jan 5;20(1):7. doi: 10.1186/s12891-018-2384-0. PMID 30611229

DOCUMENTS (1):
  • Statistical Analysis Plan: SAP NORDSTEN.DS. CEA 02.03 (2025-02-03): https://cdn.clinicaltrials.gov/large-docs/74/NCT02051374/SAP_002.pdf